CLINICAL TRIAL: NCT04229199
Title: Effectiveness of Preoperative Tour in Simulation Operating Theater in Reducing Preoperative Anxiety in Children and Their Parents: A Pragmatic, Single-blinded, Randomized Controlled Trial
Brief Title: Effectiveness of Preoperative Tour in Simulation Operating Theater in Reducing Preoperative Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Hussein A. Battah, Principal Investigator, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-534
Record Dates: First submitted 2020-01-02; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: data collectors were unaware of participants groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (IG) (Experimental): Dyads of children and parents allocated to the IG were taken into a tour to a simulation operating room accompanied by an expert anesthesia technologist two weeks before the day of surgery. This simulation operating theater is a real operating room equipped with a surgical trolley, sealing surgical lights, anesthesia machine, vital signs monitor, stethoscope, surgical trays, surgical sink, and gas supply pendent. It was prepared with popular cartoon characters, child manikin, and face masks connected to the anesthesia circuit and re-breathing bag. After being assessed by anesthesia clinic doctors, children and their parents in the IG were given a chance to visit the simulation operating room, to receive orientation, education, and demonstration orientation about what they are going to experience in the operating room. Children were encouraged to apply vital signs monitoring, and to simulate providing mask anesthesia induction to a child manikin.
  Interventions: Behavioral: simulation
- control group (CG) (No Intervention): Dyads assigned to the CG were provided only the standard practice on their day admission to the hospital.

INTERVENTIONS:
Behavioral: simulation — Dyads allocated to the IG were taken into a tour to a simulation operating room accompanied by an expert anesthesia technologist two weeks before the day of surgery. This simulation operating theater is a real operating room equipped with a surgical trolley, sealing surgical lights, anesthesia machine, vital signs monitor, stethoscope, surgical trays, surgical sink, and gas supply pendent. It was prepared with popular cartoon characters, child manikin, and face masks connected to the anesthesia circuit and re-breathing bag. After being assessed by anesthesia clinic doctors, children and their parents in the IG were given a chance to visit the simulation operating room, to receive orientation, education, and demonstration orientation about what they are going to experience in the operating room. Children were encouraged to apply vital signs monitoring, and to simulate providing mask anesthesia induction to a child manikin.
  Arms: intervention group (IG)

SUMMARY:
this study conducted to evaluate the effectiveness of preoperative tour to simulation operating theater on reducing children's and parents' preoperative anxiety. half of the participant were taken in a tour to a simulation operating theater before the day of operation and the other half were given the standard of care.

DETAILED DESCRIPTION:
the investigators examined the effectiveness of a preoperative tour to a simulation operating theater guided by an expert anesthesia technologist on reducing the Preoperative anxiety levels for children who were scheduled for elective day case procedures under general anesthesia, and their parents' anxiety levels through a 10-months randomized controlled trial at tertiary medical center in Riyadh-Saudi Arabia, and confirmed that children and parents who received the intervention had significantly lower preoperative anxiety levels than controlled children and parents.

Given that, the results showed critical levels of preoperative anxiety among school age children, and that preoperative tour to simulation operating theater as a child-friendly maneuver is directly applicable and could be considered for children scheduled for day-case procedures under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* children who were scheduled for elective day-case procedures under general anesthesia at KFMC.
* class 1 or 2 according to the American society of anesthesiology physical status.

Exclusion Criteria:

* diagnosed as having mental or psychological disorders.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
children's preoperative anxiety at holding area. | at holding area before pushing patients inside operating theater.
  measured using the modified-Yale Pre-Operative Anxiety Scale (m-YPAS). The m-YPAS is an observational anxiety scale used to assess anxiety levels in the preoperative period and during the induction of anesthesia. The total score of the scale ranged from 23 to 100, and the higher score means a worse outcome. The reference point to define high anxiety cases in the preoperative period is 30.
children's preoperative anxiety inside operating theater. | immediately before anesthesia induction.
  measured using the modified-Yale Pre-Operative Anxiety Scale (m-YPAS). The m-YPAS is an observational anxiety scale used to assess anxiety levels in the preoperative period and during the induction of anesthesia. The total score of the scale ranged from 23 to 100, and the higher score means a worse outcome. The reference point to define high anxiety cases in the preoperative period is 30.
parents' anxiety | during the procedure.
  a self-administered questionnaire, Parents' anxiety was assessed using a validated version of Beck Anxiety Inventory Scale (BAIS) into Arabic. The total scale score range from 0 to 63, where a score of 0-9 indicates no anxiety, 10-18 mild anxiety, 19-29 moderate anxiety, and 30-63 severe anxiety.
change from baseline in children's heart rate (HR) as a somatic response to anxiety | two time-points, baseline measures of HR at holding area, and secondly inside the operating theater immediately before anesthesia induction.
  somatic signs of anxiety, including children's heart rate (HR) were recorded.
change from baseline in children's systolic blood pressure (SBP) as a somatic response to anxiety | two time-points, baseline measures of SBP at holding area, and secondly inside the operating theater immediately before anesthesia induction.
  somatic signs of anxiety, including children's systolic blood pressure (SBP) were recorded.
parents' presence during anesthesia induction | at the time of anesthesia induction during the study period.
  the parents' attendance inside operating theater during anesthesia induction for their child, measured as (Yes or No).

OTHER OUTCOMES:
children's age | upon recruitment.
  the age of child participants measured by years.
children's gender | upon recruitment.
  the gender of child participants (male, female)
parent relationship status. | upon recruitment.
  the child living with (parents, mother, father, others)
history of previous anesthesia | upon recruitment.
  the child previous history of general anesthesia, measured as (Yes or No).

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Battah, MSN, Principal Investigator — King Fahad Medical City
Locations (1):
- king Fahad Medical City, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No